CLINICAL TRIAL: NCT02587819
Title: An Open-Label Phase 1 Investigation of the Safety and Tolerability of BSCT (Anti-nf-P2X7) 10% Ointment When Applied Twice Daily for 28 Days in Male and Female Patients With Basal Cell Carcinoma
Brief Title: Investigation of the Safety and Tolerability of BSCT (Anti-nf-P2X7) 10% Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosceptre (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol BSCT-001
Record Dates: First submitted 2015-10-21; First posted 2015-10-27 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Basal Cell (BCC)
MeSH Terms: conditions — Carcinoma | interventions — Therapeutics; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with BSCT (Experimental): 21 patients with BCC were treated with BSCT (anti-nf-P2X7) 10% Ointment topically applied twice daily for 28 consecutive days.
  Interventions: Drug: Treatment with BSCT

INTERVENTIONS:
Drug: Treatment with BSCT — The study product BSCT (anti-nf-P2X7) 10% Ointment was anti-nf-P2X7 (highly purified sheep IgG) in an ointment formulation for topical administration. The formulation contained 10% weight by weight of the active pharmaceutical ingredient in an anhydrous ointment base.
  Fifty (50) to 100 mg of product (an amount the size of a small pea) was applied topically twice a day for 28 days to a 25 cm2 area of skin containing a single BCC lesion. The product was to be applied in the morning and in the evening after washing.
  Other Names: BSCT (anti-nf-P2X7) 10% Ointment

SUMMARY:
This is a Phase 1, open-label, single-arm, multicenter study to assess the safety and tolerability of BSCT (anti-nf-P2X7) 10% Ointment in subjects with BCC.

DETAILED DESCRIPTION:
The purpose of the trial was to determine the safety and tolerability of BSCT (anti-nf-P2X7) 10% Ointment topically applied twice daily for 28 consecutive days in male and female patients with BCC; and to determine the steady-state pharmacokinetics (PK) of the active pharmaceutical ingredient (total sheep Immunoglobulin G [IgG]) when BSCT (anti-nf-P2X7) 10% Ointment is applied twice daily to BCC lesions. This was an open-label, single-arm, multicenter Phase 1 study that enrolled 21 BCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years of age;
* One primary histologically confirmed BCC lesion, not located on the hand or foot, suitable for surgical excision, with a minimum area of 0.5 cm2 and a maximum diameter of 2.0 cm (histological diagnosis made no more than 4 weeks prior to the Screening visit.
* Willing to refrain from using non-approved lotions or creams on the BCC treatment site and surrounding area during the treatment period and from washing the treated area for at least 8 hours following each application of study medication;
* Ability to follow study instructions and likely to complete all study requirements;
* Written informed consent obtained, including consent for biopsy tissue to be examined and stored by the central dermatopathologist;
* Written consent to allow photographs of the BCC lesion to be used as part of the study data;
* For females of childbearing potential, a negative pregnancy test at Screening and use of an acceptable form of birth control.

Exclusion Criteria:

* Pregnant, lactating, or planning pregnancy during the study;
* Presence of known or suspected systemic cancer;
* Histological evidence of squamous cell carcinoma (SCC) or any tumor other than BCC in the biopsy specimen;
* Histological evidence of severe squamous metaplasia, infiltrative, desmoplastic, or micronodular growth patterns in the biopsy specimen;
* Evidence of dermatological disease or confounding skin condition within the 25-cm2 treatment area, eg, SCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, or xeroderma pigmentosa;
* Concurrent disease or treatment that suppresses the immune system;
* Chronic medical condition that in the judgment of the investigator would interfere with the performance of the study or would place the patient at undue risk;
* Known sensitivity to any of the ingredients in the study medication;
* Treatment with systemic chemotherapeutic agents (eg, methotrexate, paclitaxel) within the 6 months prior to the Baseline visit;
* Use of systemic retinoids within the 6 months prior to the Baseline visit;
* Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the Baseline visit;
* Use of topical immunomodulators within 2 cm of the target treatment area within the 4 weeks prior to the Baseline visit;
* Treatment with topical agents for the treatment of BCC or actinic keratosis within 2 cm of the target treatment area within the 4 weeks prior to the Baseline visit:
* Treatment with liquid nitrogen, surgical excision or curettage within 2 cm of the target treatment area during the 4 weeks prior to the Baseline visit;
* Clinically significant abnormalities as noted in the screening ECG, physical examination, or laboratory test results;
* Evidence of current chronic alcohol or drug abuse which, in the investigator's opinion, might interfere with the subject's adherence to protocol requirements;
* Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the Baseline visit;
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions of the protocol and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angus Gidely-Baird, PhD, Study Director — Scientific Director - Biosceptre

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With BSCT: BSCT (anti-nf-P2X7) 10% Ointment topically applied twice daily for 28 consecutive days
Period: Overall Study
Arm/Group | Treatment With BSCT
Started | 21
Exposed | 21
Completed | 19
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With BSCT
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Adverse events and any changes in physical examinations will be monitored, as described in the Code of Federal Regulations (CFR) Title 21 Part 312. In particular local cutaneous irritation including erythema, peeling, dryness, itching, and burning/ stinging that first occur during the study or represent a worsening from Baseline will be recorded as AEs.
Time Frame: 8 weeks
Population: All (21 of 21) subjects returned for safety and tolerability assessments at days 3, 8, 15 and 29 post-Baseline. 20 of 21 patients returned for final safety assessments was at 57 days post-Baseline.
Measure: Number; unit: participants
Groups:
- Treatment With BSCT: BSCT (anti-nf-P2X7) 10% Ointment topically applied twice daily for 28 consecutive days post baseline to all subjects. All (21 of 21) subjects returned for safety and tolerability assessments at days 3, 8, 15 and 29 post-Baseline. 20 of 21 patients returned for final safety assessments at 57 days post-Baseline.
Arm/Group | Treatment With BSCT
Number analyzed (Participants) | 21
participants
  Subjects with any Serious Adverse Events | 1
  Subjects with Treatment-emergent Adverse Event(s) | 12

2. Primary Outcome: Pharmacokinetics - Measure Serum Concentration of Total Sheep IgG Using an ELISA.
Description: To determine PK, blood levels of sheep IgG were measured in samples collected at Visit 2 (Baseline), Visit 5, predose at Visit 6 (EOT), and then at 1 h, 2 h, and 4 h after the last dose of study medication.
Time Frame: 28 days
Population: At all timepoints, the serum concentration of sheep IgG was too low to be quantified in most of the subjects. One subject had measurable sheep IgG at 1 hr post dose at Visit 6 (EOT) and 3 other subjects had measurable sheep IgG at predose timepoints. In outcome measure below NA represents readings less than lower limit of quantification.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Treatment With BSCT
Number analyzed (Participants) | 21
ng/ml
  Pre-dose - Baseline visit | NA [NA to NA] — All patients had levels of sheep IgG below limit of quantitation.
  Pre dose - Visit 5 | NA [NA to 24.68] — The majority of patients had levels of sheep IgG below limit of quantitation.
  Pre dose - Visit 6 | NA [NA to 22.85] — The majority of patients had levels of sheep IgG below limit of quantitation.
  1 hour post dose - Visit 6 | NA [NA to 7.08] — The majority of patients had levels of sheep IgG below limit of quantitation.
  2 hours post dose - Visit 6 | NA [NA to NA] — All patients had levels of sheep IgG below limit of quantitation.
  4 hours post dose - Visit 6 | NA [NA to NA] — All patients had levels of sheep IgG below limit of quantitation.

3. Primary Outcome: Pharmacokinetics - Measure Subject Antibody Response to the Active Pharmaceutical Ingredient Using an Indirect Fluorescent Immuno Assay.
Description: The active ingredient of BSCT is sheep IgG which may causes an immunogenic response if it enters the systemic circulation. To monitor this response patient blood samples collected at Screening, Visit 2 (Baseline), Visit 6 (EOT), and at Visit 8 (EOS) was tested for anti-sheep IgG antibodies (indicative of immune response against API).
Time Frame: 8 weeks
Population: Anti sheep IgG antibody titres were measured from 21 subjects at screening and baseline, 20 subjects at Visit 6 (Day 29 EOT) and 19 subjects at Visit 8 (Day 57 follow up). The percentage of patients with detectable anti sheep antibodies is reported.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment With BSCT
Number analyzed (Participants) | 21
percentage of subjects
  Subjects with anti sheep IgG at screening | 42.9
  Subjects with anti sheep IgG at Baseline | 38.1
  Subjects with anti sheep IgG at visit 6 | 50
  Subjects with anti sheep IgG at visit 8 | 52.6

4. Post Hoc Outcome: Change in Lesion Size.
Description: BCC lesion area was measured at Baseline and after 28 days treatment. Percantage change in lesion area was caculated.
Time Frame: 28 days
Population: Final area of lesion was not recorded for one subject.
Measure: Mean (Standard Error); unit: percentage change in tumour area
Arm/Group | Treatment With BSCT
Number analyzed (Participants) | 20
percentage change in tumour area | -12.86 (5.88)

ADVERSE EVENTS:
Time Frame: 8 weeks (28 day treatment period and 28 day follow up period).
Description: All (21 of 21) subjects returned for safety and tolerability assessments at days 3, 8, 15 and 29 post-Baseline. 20 of 21 patients returned for final safety assessments was at 57 days post-Baseline.
Arm/Group | Treatment With BSCT
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With BSCT (N=21)
Acute myocardial infarction (Cardiac disorders) | 1 (1) — Subject 01-007 experienced a myocardial infarction from 9 September 2013 (Study Day 49) to 11 September 2013 (Study Day 51), which was moderate and was considered to be unrelated to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With BSCT (N=21)
Application site dryness (General disorders) | 7 (7)
Application site erythema (General disorders) | 10 (10)
Application site exfoliation (General disorders) | 5 (5)
Application site pain (General disorders) | 3 (3)
Application site pruritus (General disorders) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No